CLINICAL TRIAL: NCT04508387
Title: The Effects of CO2 Pneumoperitoneum at Different Temperature and Humidity on Hemodynamic and Respiratory Parameters and Postoperative Pain in Gynecological Laparoscopic Surgery: A Prospective Randomized Controlled Study
Brief Title: The Effects of CO2 Pneumoperitoneum at Different Temperature in Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, asuman özdemir, doctor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EGE19-3.1/40
Record Dates: First submitted 2020-07-14; First posted 2020-08-11 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Benign Neoplasm of Cervix Uteri; Gynecological Laparoscopy
Keywords: Gynecological laparoscopy; standard CO2; heated-humidified CO2; hemodynamic parameters; respiratory parameters

STUDY DESIGN:
Intervention Model Description: The patients were divided into two groups according to a randomization scheme created by a computer: Group CD (cold-dry) patients were administered dry CO2 via insufflator at room temperature (21°C), while Group HH (heated-humidified) patients were administered 95% humidified CO2 insufflation at 37°C. The study was planned as a randomized and double-blind study, where patients were not informed of their group. During the operation and in the postoperative period, the patients were followed up by two different anesthetists. All patients were given information and training on the anesthesia method, the use of the patient-controlled-analgesia (PCA) device and the visual analog scale (VAS) the day before the operation. The patients' demographic data (age, weight, height, etc.) and their basal systolic, diastolic and mean blood pressures and heart rates were measured prior to the operation and recorded on the case report form.
Who Masked: Investigator
Masking Description: The study was planned as a randomized and double-blind study, where patients were not informed of their group. During the operation and in the postoperative period, the patients were followed up by two different anesthetists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group HH (heated-humidified) patients (Active Comparator): Group HH (heated-humidified) patients were administered 95% humidified CO2 insufflation at 37°C. All patients were given information and training on the anesthesia method, the use of the patient-controlled-analgesia (PCA) device and the visual analog scale (VAS) the day before the operation. The patients' demographic data (age, weight, height, etc.) and their basal systolic, diastolic and mean blood pressures and heart rates were measured prior to the operation and recorded on the case report form.
  Interventions: Procedure: Group HH (heated-humidified)
- Group CD (cold-dry) patients (Placebo Comparator): Group CD (cold-dry) patients were administered dry CO2 via insufflator at room temperature (21°C). All patients were given information and training on the anesthesia method, the use of the patient-controlled-analgesia (PCA) device and the visual analog scale (VAS) the day before the operation. The patients' demographic data (age, weight, height, etc.) and their basal systolic, diastolic and mean blood pressures and heart rates were measured prior to the operation and recorded on the case report form.
  Interventions: Procedure: Group HH (heated-humidified)

INTERVENTIONS:
Procedure: Group HH (heated-humidified) — Group CD patients were administered dry CO2 via insufflator at room temperature (21°C), while Group HH patients were administered 95% humidified CO2 insufflation at 37°C. The study was planned as a randomized and double-blind study, where patients were not informed of their group. During the operation and in the postoperative period, the patients were followed up by two different anesthetists. All patients were given information and training on the anesthesia method, the use of the patient-controlled-analgesia device and the visual analog scale the day before the operation. The patients' demographic data (age, weight, height, etc.) and their basal systolic, diastolic and mean blood pressures and heart rates were measured prior to the operation and recorded on the case report form. Both groups received the standard general anesthesia protocol. Laparoscopic surgery was performed in the same manner for all cases by AA.

SUMMARY:
Objective: It is recommended to heat and humidify CO2 in laparoscopic surgery to prevent postoperative pain and hypothermia but information about its effects on hemodynamic and respiratory parameters is limited. The investigators aimed to investigate the effects of standard and heated-humidified CO2 on hemodynamic and respiratory parameters.

Study design: One hundred patients who underwent laparoscopic hysterectomy for benign pathology were divided into two groups: Group CD (cold-dry) patients were administered standard CO2, while Group HH (heated-humidified) patients were administered 95% humidified insufflation at 37°C. Hemodynamic and respiratory parameters, body temperature, pain score and blood count parameters were recorded.

DETAILED DESCRIPTION:
The sample consisted of 100 American Society of Anesthesiologists (ASA) physical status I-II patients aged 40-65 who underwent laparoscopic hysterectomy for benign pathology. The patients were divided into two groups according to a randomization scheme created by a computer: Group CD (cold-dry) patients were administered dry CO2 via insufflator at room temperature (21°C), while Group HH (heated-humidified) patients were administered 95% humidified CO2 insufflation at 37°C. The study was planned as a randomized and double-blind study, where patients were not informed of their group.During the operation and in the postoperative period, the patients were followed up by two different anesthetists. All patients were given information and training on the anesthesia method, the use of the patient-controlled-analgesia (PCA) device and the visual analog scale (VAS) the day before the operation. The patients' demographic data (age, weight, height, etc.) and their basal systolic, diastolic and mean blood pressures and heart rates were measured prior to the operation and recorded on the case report form.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II patients aged 40-65 who underwent laparoscopic hysterectomy for benign pathology.

Exclusion Criteria:

* Patients with chronic obstructive pulmonary disease, asthma, advanced liver and kidney disease, infection, bleeding disorder and drug allergies

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
hemodynamic parameters: diastolic and mean blood pressure | In the operation period
  diastolic and mean blood pressure
body temperature | In the operation period
  body temperature
respiratory parameters: tidal volume | In the operation period
  tidal volume

SECONDARY OUTCOMES:
Visual Analogue Scale | 24 hour
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'.(VAS:0 no pain, VAS:10 very severe pain)
morphine consumption | 24 hour
  pain

CONTACTS AND LOCATIONS:
Overall Officials: Ilkben gunusen, 1, Study Director — Ege University
Locations (1):
- Asuman Sargin, Izmir, Anesthesiology and Reanimation, Ege Uni, Turkey (Türkiye)

REFERENCES:
- [Background] Scott JE, Singh A, Valverde A, Blois SL, Foster RA, Kilkenny JJ, Linden AZ. Effect of pneumoperitoneum with warmed humidified or standard-temperature carbon dioxide during laparoscopy on core body temperature, cardiorespiratory and thromboelastography variables, systemic inflammation, peritoneal response, and signs of postoperative pain in healthy mature dogs. Am J Vet Res. 2018 Dec;79(12):1321-1334. doi: 10.2460/ajvr.79.12.1321. PMID 30457909
- [Result] Birch DW, Dang JT, Switzer NJ, Manouchehri N, Shi X, Hadi G, Karmali S. Heated insufflation with or without humidification for laparoscopic abdominal surgery. Cochrane Database Syst Rev. 2016 Oct 19;10(10):CD007821. doi: 10.1002/14651858.CD007821.pub3. PMID 27760282
- [Result] Cheong JY, Keshava A, Witting P, Young CJ. Effects of Intraoperative Insufflation With Warmed, Humidified CO2 during Abdominal Surgery: A Review. Ann Coloproctol. 2018 Jun;34(3):125-137. doi: 10.3393/ac.2017.09.26. Epub 2018 Jun 30. PMID 29991201
- [Derived] Gunusen I, Akdemir A, Sargin A, Karaman S. The effects of CO2 pneumoperitoneum at different temperature and humidity on hemodynamic and respiratory parameters and postoperative pain in gynecological laparoscopic surgery: A prospective randomized controlled study. Asian J Surg. 2022 Jan;45(1):154-161. doi: 10.1016/j.asjsur.2021.04.005. Epub 2021 Apr 20. PMID 33888367

DOCUMENTS (1):
  • Study Protocol (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT04508387/Prot_002.pdf